CLINICAL TRIAL: NCT03936465
Title: Phase 1 Study of the Bromodomain (BRD) and Extra-Terminal Domain (BET) Inhibitors BMS-986158 and BMS-986378 (CC-90010) in Pediatric Cancer
Brief Title: Study of the Bromodomain (BRD) and Extra-Terminal Domain (BET) Inhibitors BMS-986158 and BMS-986378 in Pediatric Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Stand Up To Cancer (Other)
Responsible Party: Principal Investigator, Steven DuBois, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-040
Record Dates: First submitted 2019-04-30; First posted 2019-05-03 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumor, Childhood; Lymphoma; Brain Tumor, Pediatric
Keywords: Solid Tumor; Lymphoma; Neuroblastoma; Sarcoma; Medulloblastoma; MYC; MYCN; BRD4; BET inhibitor; Bromodomain
MeSH Terms: conditions — Lymphoma; Brain Neoplasms; Neuroblastoma; Sarcoma; Medulloblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 Cohort A (Experimental): * Patients will receive BMS-986158 monotherapy orally for 5 days on / 2 days off per week in 28-day cycles.
  * Patients with unselected relapsed or refractory solid tumors or lymphoma
  Interventions: Drug: BMS-986158
- Arm 1 Cohort B (Experimental): * Patients will receive BMS-986158 monotherapy orally for 5 days on / 2 days off per week in 28-day cycles.
  * Patients with relapsed or refractory solid tumors or lymphoma that have defined molecular features predicted to increase sensitivity to BET inhibition
  Interventions: Drug: BMS-986158
- Arm 2 Cohort A (Experimental): * Patients will receive BMS-986378 (also known as CC-90010) monotherapy orally for 4 days every 28 days.
  * Patients with relapsed or refractory CNS tumors or CNS metastatic tumors
  Interventions: Drug: BMS-986378
- Arm 2 Cohort B (Experimental): * Patients will receive BMS-986378 (also known as CC-90010) monotherapy orally for 4 days every 28 days.
  * Patients with relapsed or refractory CNS tumors or CNS metastatic tumors that have defined molecular features predicted to increase sensitivity to BET inhibition
  Interventions: Drug: BMS-986378

INTERVENTIONS:
Drug: BMS-986158 — BMS-986158 belongs to a group of drugs called Bromodomain (BRD) and Extra-Terminal Domain (BET) inhibitors. These drugs block proteins that are important in reading DNA, which is a process important for cancer cells.
  Arms: Arm 1 Cohort A; Arm 1 Cohort B
Drug: BMS-986378 — BMS-986378 (also known as CC-90010) belongs to a group of drugs called Bromodomain (BRD) and Extra-Terminal Domain (BET) inhibitors. These drugs block proteins that are important in reading DNA, which is a process important for cancer cells.
  Other Names: CC-90010
  Arms: Arm 2 Cohort A; Arm 2 Cohort B

SUMMARY:
Arm 1 of this research study is studying an investigational drug called BMS-986158 as a possible treatment for pediatric solid tumors or lymphoma. Arm 2 of this research study is studying an investigational drug called BMS-986378 (also known as CC-90010) as a possible treatment for pediatric brain tumors or pediatric tumors that have spread to the brain.

DETAILED DESCRIPTION:
This is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved BMS-986158 or BMS-986378 as a treatment for any disease.

BMS-986158 and BMS-986378 are currently still being studied in adults. This is the first time that BMS-986158 or BMS-986378 will be evaluated in younger children, though children 12-17 years of age may also be included in parts of adult studies of BMS-986158.

Research in the laboratory has shown that BMS-986158 and BMS-986378 may have activity against cancer cells. These drugs belong to a group of drugs called Bromodomain (BRD) and Extra-Terminal Domain (BET) inhibitors. These drugs block proteins that are important in reading DNA, which is a process important for cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 21 years at time of enrollment. Note the requirement in section 3.1.6 that all patients must be able to swallow intact capsules.
* Karnofsky performance status ≥ 50% for patients ≥16 years of age or Lansky ≥ 50% for patients <16 years of age (see Appendix A)
* Diagnosis requirement

  * Participants must have evaluable or measurable disease (see Section 11).
  * Must have disease that is relapsed or refractory and for which standard curative measures do not exist or are no longer effective.
  * For Arm 1, Cohort 1A, participants must have histologically confirmed non-CNS primary solid tumors or lymphoma based upon biopsy or surgery at relapse/progression. Patients without biopsy or surgery at relapse/progression and with tissue only available from initial diagnosis may still be considered after discussion with the overall Primary Investigator.
  * For Arm 1, Cohort 1B, participants must have histologically confirmed solid tumors or lymphoma based upon biopsy or surgery at relapse/progression as well as documentation of one of the following confirmed tumor molecular features obtained in a laboratory certified to return results for clinical purposes. Patients without biopsy or surgery at relapse/progression and with tissue only available from initial diagnosis may still be considered after discussion with the overall Primary Investigator.
  * MYCN amplification or high copy number gain
  * MYC amplification or high copy number gain
  * Translocation involving MYC or MYCN
  * Translocation involving BRD4 or BRD3
  * BRD4 amplification or high copy number gain
  * Histologic diagnosis of NUT midline carcinoma
  * For Arm 2, Cohort 2A, participants must have histologically confirmed primary CNS p tumors or untreated CNS metastases based upon biopsy or surgery at relapse/progression. Patients without biopsy or surgery at relapse/progression and with tissue only available from initial diagnosis may still be considered after discussion with the overall Primary Investigator.
  * For Arm 2, Cohort 2B, participants must have histologically confirmed primary CNS p tumors or untreated CNS metastases based upon biopsy or surgery at relapse/progression as well as documentation of one of the following confirmed tumor molecular features obtained in a laboratory certified to return results for clinical purposes. Patients without biopsy or surgery at relapse/progression and with tissue only available from initial diagnosis may still be considered after discussion with the overall Primary Investigator.
  * MYCN amplification or high copy number gain
  * MYC amplification or high copy number gain
  * Translocation involving MYC or MYCN
  * Translocation involving BRD4 or BRD3
  * BRD4 amplification or high copy number gain
  * Histologic diagnosis of NUT midline carcinoma
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy except organ function as noted in Section 3.1.5. Patients must meet the following minimum washout periods prior to enrollment:
* Myelosuppressive chemotherapy: At least 21 days after the last dose of myelosuppressive chemotherapy (42 days for nitrosourea or mitomycin C).
* Radiotherapy:

  * At least 14 days after local XRT (small port, including cranial radiation);
  * At least 90 days must have elapsed after prior TBI, or if >50% radiation of pelvis;
  * At least 180 days must have elapsed after prior craniospinal XRT;
  * At least 42 days must have elapsed if other substantial BM radiation;
  * At least 42 days must have passed since last MIBG or other radionuclide therapy.
* Small molecule biologic therapy: At least 7 days following the last dose of a small molecule biologic agent. For agents with known adverse events occurring beyond 7 days, this duration must be extended beyond the time in which adverse events are known to occur. If extended duration is required, this must be discussed with and approved by the overall PI.
* Monoclonal antibody: At least 28 days must have elapsed after the last dose of therapeutic monoclonal antibody.
* Myeloid growth factors: At least 14 days following the last dose of long-acting growth factor (e.g. Neulasta) or 7 days following short-acting growth factor.
* Autologous hematopoietic stem cell transplant and stem cell boost: Patients must be at least 60 days from day 0 of an autologous stem cell transplant or autologous stem cell boost.
* Cellular therapies (including CAR-T cells) and other non-cellular, non-antibody immunotherapies (e.g., vaccines): At least 42 days must have elapsed after last dose.
* Major Surgery: At least 2 weeks from prior major surgical procedure. Note: Major surgical procedure will be considered all surgical procedures aside from the following: Biopsy; central line placement/removal; bone marrow aspirate/biopsy; lumbar puncture; dental procedures; gastrostomy tube placement; and VP shunt placement/revision.
* BET inhibitors: Patients must not have received prior treatment with a BET inhibitor, except patients with CNS tumors or CNS metastasis previously treated on Arm 1 of the trial who discontinued protocol therapy due to disease progression and not due to toxicity. Such patients may participate in Arm 2 of the trial.
* Participants must have normal organ function as defined below.
* Bone Marrow Function
* For Patients without Documented Bone Marrow Involvement by Disease:

  * Hemoglobin > 8 g/dL (may be transfused)
  * Absolute neutrophil count ≥ 1,000 /uL
  * Platelets ≥ 100,000 /uL and transfusion independent, defined as not receiving a platelet transfusion for at least 5 days prior to CBC documenting eligibility.
* For Patients with Documented Bone Marrow Involvement by Disease:

  * Hemoglobin > 8 g/dL (may be transfused)
  * Absolute neutrophil count ≥ 750 /uL
  * Platelets ≥ 75,000 /uL and transfusion independent, defined as not receiving a platelet transfusion for at least 5 days prior to CBC documenting eligibility.
* Hepatic Function:

  * Total bilirubin ≤ 1.5 x upper limit of normal for age (patients with known Gilbert's may be considered after discussion with overall PI and if direct bilirubin is at or below the upper limit of normal for age)
  * ALT (SGPT) ≤ 3 x upper limit of normal (135 U/L) For the purpose of this study, the ULN for ALT is 45 U/L
  * Serum albumin > 2 g/dL
* Adequate Pancreatic Function:

  --Lipase < upper limit of normal
* Adequate GI Function:

  --Diarrhea < grade 1 by CTCAE version 5
* Coagulation Factors:

  * International Normalized Ratio (INR) < 1.5
  * Partial thromboplastin time (PTT) < 1.5 times upper limit of normal
* For patients having labs drawn via heparinized catheters, it is important to request heparin-absorbed values.
* Adequate Cardiac Function:

  --QTc < 480 msec
* Renal Function:

  * A serum creatinine within protocol limits based on age/sex.

OR

* Creatinine clearance ≥ 60 mL/min/1.73 m2 for participants with creatinine levels greater than the above age/sex maximum allowed values.
* Able to swallow intact capsules (BMS-986158) or tablets (BMS-986378, also known as CC-90010).
* Patient (or parent or legally authorized representative, if minor) is able to understand and willing to provide informed consent, using an institutionally approved informed consent procedure.
* Participants of childbearing or child-fathering potential must agree to use adequate contraception throughout their participation following the guidance in Appendix H.

Exclusion Criteria:

* Prior solid organ or allogeneic stem cell transplantation.
* Patients with primary or metastatic CNS tumors are not eligible for Arm 1, except:

  --Patients with a history of CNS metastatic disease that has been resected and/or radiated without evidence of active CNS disease for 3 months preceding enrollment; NOTE: patients with primary CNS tumors or solid tumors with active CNS metastases will be eligible for Arm 2.
* Patients receiving any of the following prohibited foods and medications:

  * Agents listed in Appendix B within 7 days prior to enrollment
  * Grapefruit or Seville oranges and/or their juices within 7 days prior to enrollment
  * Non-steroidal anti-inflammatory drugs, oral anticoagulants, and therapeutic heparins (unfractionated or low molecular weight heparin) at the time of enrollment. Note: Use of heparin to maintain patency of a central or peripheral catheter is allowed
  * Other investigational agents being administered under an IND.
* Pregnant participants will not be entered on this study given that the effects of BMS-986158 and BMS-986378 (CC-90010) on the developing human fetus are unknown. Female participants of childbearing potential must have a documented negative pregnancy exam within 24 hours prior to dosing.
* Breastfeeding mothers are not eligible, because there is an unknown risk for adverse events in nursing infants secondary to treatment of the mother with BMS-986158 or BMS-986378 (CC-90010).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to BMS-986158 or BMS-986378 (CC-90010).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with a known history of HIV, hepatitis B, and/or hepatitis C (testing not required as part of screening).
* Patients with gastrointestinal disease or disorder that could interfere with absorption of BMS-986158 or BMS-986378 (CC-90010), such as bowel obstruction or inflammatory bowel disease.
* For Arm 1: Patients with BSA < 0.3 m2 for all dose levels except Dose Level -2 or -2i for which patients with BSA < 0.71 m2 will be excluded due to dose rounding constraints.
* For Arm 2: Patients with BSA < 0.65 m2.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity Rate | 28 days (first cycle)
  Dose limiting toxicity as defined in protocol
The Rate of Toxicities from Protocol Therapy | 2 years
  Adverse events coded using CTCAE version 5

SECONDARY OUTCOMES:
Objective Response Rate | 2 years
  Objective response rate
Pharmacokinetics of BMS-986158 (Arm 1) or BMS-986378 (Arm 2) | 2 years
  Plasma concentrations of BMS-986158 or BMS-986378
Pharmacodynamics of BMS-986158 (Arm 1) or BMS-986378 (Arm 2) | 2 years
  Gene expression levels in peripheral blood
Blood Markers of Response | 2 years
  Levels of ctDNA in peripheral blood
CSF Markers of Response | 2 years
  Levels of ctDNA in CSF
Tumor Markers of Response | 2 years
  Levels of Myc proteins in tumor

CONTACTS AND LOCATIONS:
Overall Officials: Steven G. DuBois, MD, MS, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (5):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Seattle Children's Hospital, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No